CLINICAL TRIAL: NCT04878952
Title: Activity Monitoring to Improve Patient Care During Chemoradiotherapy for Locally Advanced Non-Small Cell Lung Cancer (LA-NSCLC)
Brief Title: Testing the Addition of Activity Monitoring With a Wearable Electronic Device to Improve Patient Care During Treatment for Lung Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: will not be able to meet study accrual objectives.
Sponsor: NRG Oncology (Other)
Collaborators: Pennsylvania Department of Health Commonwealth Universal Research Enhancement Program (PA CURE) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NRGF-001
Record Dates: First submitted 2021-04-30; First posted 2021-05-10 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Non-small Cell Lung Cancer; Non-small Cell Lung Cancer Stage III; Recurrent Non Small Cell Lung Cancer
Keywords: Locally advanced non-small cell lung cancer; LA-NSCLC; Activity Tracking
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I: Usual Care (No Intervention): Patients will receive their usual care of thoracic radiotherapy with concurrent chemotherapy.
- Arm II: Usual Care + Continuous physical activity monitoring via a wearable device (Experimental): Patients will receive their usual care of thoracic radiotherapy with concurrent chemotherapy along with continuous physical activity monitoring via a wearable device.
  Interventions: Other: Garmin Vivofit Activity Tracker

INTERVENTIONS:
Other: Garmin Vivofit Activity Tracker — Activity tracker that is worn on the wrist.
  Arms: Arm II: Usual Care + Continuous physical activity monitoring via a wearable device

SUMMARY:
This trial will examine if the monitoring of daily step counts during a course of concurrent chemoradiotherapy for locally advanced non-small cell lung cancer will enable clinicians to deliver improved supportive care and reduce the rate of adverse events during the course of radiation treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To demonstrate that monitoring daily step counts during a course of concurrent chemoradiotherapy for locally advanced non-small cell lung cancer will enable clinicians to deliver improved supportive care and reduce the rate of adverse clinical events during the radiotherapy course.

SECONDARY OBJECTIVES:

I. To demonstrate the feasibility of monitoring daily step counts during a course of chemoradiotherapy in the setting of a multi-institutional trial.

II. To examine the association between baseline activity level and clinical outcomes related to treatment tolerance, quality of life, chemoradiotherapy adverse events, and physical function preservation.

III. To demonstrate associations between daily step counts and short-term hospitalization risk.

IV. To explore predictors of step count decline during chemoradiotherapy among clinical factors and radiotherapy plan parameters.

EXPLORATORY OBJECTIVES:

I. To explore patterns of care regarding adjuvant immunotherapy administration following definitive chemoradiotherapy for locally advanced non-small cell lung cancer.

II. To examine the association between baseline activity level with progression free survival and overall survival.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Usual Care

ARM II: Usual Care + Continuous physical activity monitoring via a wearable device.

Patients randomized to undergo activity monitoring will use a wearable device from the time of study enrollment until four weeks after the completion of thoracic radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of NSCLC
* Planned initiation (within the 30 days after study registration) of fractionated (≥15 treatments) thoracic radiotherapy with concurrent chemotherapy. Expected treatment scenarios include:

  * Definitive treatment of stage III disease (most common)
  * Definitive treatment for locoregional recurrence of early stage disease
  * Definitive treatment of unresectable stage II disease
  * Preoperative treatment of stage III disease
  * Postoperative treatment after incomplete resection (uncommon)
  * Radical treatment for a patient with advanced/metastatic disease with the goal of achieving long-term thoracic disease control (e.g., oligometastatic disease where metastases are addressed with resection or stereotactic radiotherapy)
* ECOG Performance Status 0-3 within 30 days prior to registration
* Age ≥ 18
* Ambulates independently or with a cane (use of a walker not permitted)
* Patients who already use wearable devices and/or smartphones that monitor physical activity are eligible for this trial. Patients must agree to wear the device provided by the study.
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry.

Exclusion Criteria:

* Patients with a history of another cancer that is expected to affect the toxicity profile of thoracic chemoradiotherapy for NSCLC
* Patients receiving concurrent treatment for another cancer that is expected to affect the toxicity profile of thoracic chemoradiotherapy
* Patients receiving thoracic radiotherapy without concurrent chemotherapy are ineligible. Patients receiving concurrent chemotherapy and another form of systemic therapy (e.g., immunotherapy) are eligible. Patients receiving radiotherapy with concurrent immunotherapy or targeted therapy but without chemotherapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of hospital admission | From study enrollment to 1 month after radiotherapy completion.
  Occurrence of hospital admission during radiation treatment or within 1 month after radiotherapy completion.
Occurrence of emergency room visit lasting more than 24 hours | From study enrollment to 1 month after radiotherapy completion.
  Occurrence of emergency room visit lasting more than 24 hours during radiation treatment or within 1 month after radiotherapy completion.
Occurrence of radiation treatment interruption | From study enrollment to radiotherapy completion.
  Occurrence of of radiation treatment interruption (missing two or more treatments, not due to machine issues or scheduled holidays) during radiation treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Ohri, MD, Principal Investigator — NRG Oncology
Locations (5):
- United States (5):
  - WellSpan Health - Chambersburg, Chambersburg, Pennsylvania
  - WellSpan Health - Ephrata, Ephrata, Pennsylvania
  - WellSpan Health - Gettysburg, Gettysburg, Pennsylvania
  - WellSpan Health - Lebanon, Lebanon, Pennsylvania
  - WellSpan Health - York, York, Pennsylvania